CLINICAL TRIAL: NCT01781949
Title: Effectiveness of Rapid HIV Screening Methods in Urban Emergency Departments
Brief Title: The HIV Testing Using Enhanced Screening Techniques in Emergency Departments Trial
Acronym: HIV TESTED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Denver Health and Hospital Authority (Other)
Collaborators: Alameda County Medical Center (Other); Johns Hopkins University (Other); University of Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: NIAID R01 AI106057
Record Dates: First submitted 2013-01-11; First posted 2013-02-01 (Estimated); Last update posted 2024-03-04 (Actual); Status verified 2018-09

CONDITIONS: Rapid HIV Screening
Keywords: HIV infection; Targeted screening; Nontargeted screening; Emergency department; Urgent care; Effectiveness
MeSH Terms: conditions — HIV Infections; Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- A: Nontargeted rapid HIV screening (Other): Eligible patients randomized to this arm will be offered rapid HIV screening without assessment of risk. HIV testing will occur on a 24-hour basis as part of routine ED care.
  Interventions: Other: A: Nontargeted rapid HIV screening
- B: Enhanced targeted rapid HIV screening (Other): Eligible patients randomized to this arm will be asked to answer questions regarding HIV risk using the Denver HIV Risk Score (DHRS), an empirically-developed clinical prediction instrument for assessing HIV risk, to identify patients at increased risk for HIV infection. Patients identified as being at increased risk for HIV infection will be offered rapid HIV testing. HIV testing will occur on a 24-hour basis as part of routine ED care.
  Interventions: Other: B: Enhanced targeted rapid HIV screening
- C: Traditional targeted rapid HIV screening (Other): Eligible patients randomized to this arm will be asked to answer questions related to HIV risk using a traditional behavioral risk screening tool to identify patients at increased risk for HIV infection. Patients identified as being at increased risk for HIV infection will be offered rapid HIV testing. HIV testing will occur on a 24-hour basis as part of routine ED care.
  Interventions: Other: C: Traditional targeted rapid HIV screening

INTERVENTIONS:
Other: A: Nontargeted rapid HIV screening — Patients who present to the ED for evaluation, who meet criteria for inclusion, and who are randomized to this arm will be offered voluntary, free, and confidential rapid HIV testing by nurses using opt-out consent during medical screening.
  Arms: A: Nontargeted rapid HIV screening
Other: B: Enhanced targeted rapid HIV screening — Patients who present to the ED for evaluation, who meet criteria for inclusion, and who are randomized to this arm will be asked questions from the Denver HIV Risk Score (DHRS). Patients will be considered at increased risk for HIV infection if they have a DHRS score of 30 or more. These increased-risk patients will be offered rapid HIV testing using opt-out consent by nurses during medical screening. Patients identified as low risk (DHRS <30) will not be offered rapid HIV testing but will eligible for diagnostic HIV testing.
  Arms: B: Enhanced targeted rapid HIV screening
Other: C: Traditional targeted rapid HIV screening — Patients who present to the ED for evaluation, who meet criteria for inclusion, and who are randomized to this arm will be asked questions from a Behavioral Risk Screening Tool (BRST). The BRST was adopted from the 2001 Centers for Disease Control and Prevention's recommendations for targeted HIV screening, and includes 6 questions. An affirmative response to 1 or more questions identifies the person as being at increased risk for HIV infection. These patients will be offered rapid HIV testing using opt-out consent by nurses during medical screening. Patients who do not respond affirmatively to any of the questions will not be offered rapid HIV testing but will eligible for diagnostic HIV testing.
  Arms: C: Traditional targeted rapid HIV screening

SUMMARY:
The purpose of this study is to evaluate the effectiveness of 3 modern rapid HIV screening methods, including a novel targeted strategy, in urban emergency department settings in the United States.

DETAILED DESCRIPTION:
Early identification of undiagnosed HIV infection remains a critical public health priority. In the United States, approximately 250,000 HIV-infected individuals remain undiagnosed and 50,000 new infections occur annually, despite several substantial HIV-related public health initiatives. Although HIV testing is an important intervention, controversy still exists as to how it should be implemented.

In 2006, the Centers for Disease Control and Prevention (CDC) recommended nontargeted opt-out HIV screening in clinical settings where the undiagnosed prevalence was ≥0.1%. Emergency departments (EDs) have been a major focus of these recommendations, prompted by the fact that over 120 million ED visits occur annually in the United States, they serve large proportions of underserved patients, and are the most common site of missed diagnostic opportunities for HIV infection. In contrast, in 2007 the United States Preventive Services Task Force recommended targeted HIV screening (i.e., testing high-risk subpopulations) as the principal approach to HIV testing because insufficient evidence existed to support the CDC recommendations.

Led by Jason Haukoos, MD, MSc, the research team has pioneered investigations in this area since 2004, recently publishing the largest clinical trial to date, concluding that nontargeted opt-out rapid HIV screening in the ED was associated with a small increase in number of newly-identified HIV-infected patients when compared to diagnostic testing (i.e., testing based on clinical signs or symptoms) by physicians. The investigators also recently developed the Denver HIV Risk Score (DHRS), the first multivariable tool to estimate risk of HIV infection. The DHRS combines 3 demographic and 5 behavioral characteristics, and classifies patients into distinct strata with increasing HIV prevalence.

To build on this work, the investigators propose the following specific aims: (1) to evaluate and compare the effectiveness of 3 rapid HIV screening strategies when fully-integrated into ED care; (2) to measure and compare programmatic costs of each HIV screening strategy; and (3) to measure and compare ED operational processes of each HIV screening strategy. In doing so, the investigators will perform a multi-center prospective randomized control trial to test the following hypotheses: (1) targeted rapid HIV screening using the DHRS to identify high-risk patients is significantly associated with new HIV diagnoses when compared to traditional targeted rapid HIV screening and nontargeted rapid HIV screening; (2) enhanced and traditional targeted rapid HIV screening is more cost effective per newly-identified patient than nontargeted rapid HIV screening; and (3) enhanced targeted rapid HIV screening is associated with non-inferior ED process metrics and crowding when compared to traditional targeted screening or nontargeted screening.

To accomplish these aims, the investigative team will conduct: (1) a prospective randomized controlled "pragmatic" clinical effectiveness trial in the EDs at Denver Health Medical Center (Denver, CO), Alameda County Medical Center (Oakland, CA), Johns Hopkins Hospital (Baltimore, MD), and the University of Cincinnati Medical Center (Cincinnati, OH); and (2) nested observational studies to evaluate programmatic costs and operational metrics between the 3 rapid HIV screening strategies and using newly-diagnosed HIV infection as the primary outcome.

ELIGIBILITY:
Inclusion Criteria:

* Greater than or equal to 16 years of age
* Clinically stable
* Capable of providing consent for medical care

Exclusion Criteria:

* < 16 years old
* Unable to consent for medical care
* Prisoners or detainees
* Self-identified as infected with HIV
* Occupational exposure
* Sexual assault
* Fast-track patients

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 76235 (Actual)
Dates: Start 2014-04; Primary Completion 2016-01 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Confirmed Newly-Diagnosed HIV Infection | Day 1
  Confirmed newly-diagnosed and previously-diagnosed HIV infection; classified as binary "yes" or "no"; assessed using structured medical record and laboratory data abstraction.

SECONDARY OUTCOMES:
CD4 Count | Day 1
  CD4 count (cells/mm3) at the time of diagnosis; assessed using structured laboratory data abstraction.
HIV Viral Load | Day 1
  HIV viral load (copies/mL) at the time of diagnosis; assessed using structured laboratory data abstraction.
Linkage-to-Care | Expected average of 1 week, but may be up to 1 month
  Determined by completion of a follow-up linkage-to-care visit within 30 days of initial ED diagnosis; classified as binary "yes" or "no"; assessed using structured medical record abstraction.
Development of AIDS | 1 year after diagnosis
  Using conventional definitions for the development of AIDS during any time during the year following diagnosis; classified as binary "yes" or "no"; assessed using structured medical record abstraction.
Initiation of Antiretroviral Therapy | 1 year after diagnosis
  Whether antiretroviral therapy (ART) was planned or initiated at any time during the year following diagnosis; classified as binary "yes" or "no"; assessed using structured medical record abstraction.
Treatment for Opportunistic Infections | 1 year after diagnosis
  Whether treatment for specific opportunistic infections were initiated at any time during the year following diagnosis; assessed using structured medical record abstraction.
Hospitalization | 1 year after diagnosis
  Hospitalization is defined as any unscheduled hospital admission, occurring at any time during the year following diagnosis; measured as binary "yes" or "no" and as number of unique hospitalizations; assessed using structured medical record abstraction.
Scheduled Medical Care Visits | 1 year after diagnosis
  Scheduled medical care visits is defined as all scheduled visits (both outpatient and inpatient), occurring at any time during the year following diagnosis; classified as an interval value of unique visits; assessed using structured medical record abstraction.
Unscheduled Medical Care Visits | 1 year after diagnosis
  Unscheduled medical care visits is defined as all unscheduled visits (both outpatient and inpatient), occurring at any time during the year following diagnosis; classified as an interval value of unique visits; assessed using structured medical record abstraction.
Mortality | 1 year after diagnosis
  Mortality is defined as death at any time during the year following diagnosis; classified as binary "yes" or "no"; assessed using structured medical record abstraction.

CONTACTS AND LOCATIONS:
Overall Officials: Jason S Haukoos, MD, MSc, Principal Investigator — Denver Health and Hospital Authority
Locations (4):
- United States (4):
  - Alameda County Medical Center, Oakland, California
  - Denver Health and Hospital Authority, Denver, Colorado
  - Johns Hopkins University, Baltimore, Maryland
  - University of Cincinnati Medical Center, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: Yes
The final research dataset resulting from this project will be made available to other investigators who wish to perform secondary analyses in this content area. The final dataset will include demographic and self-reported behavioral risk information as collected as a part of the Denver HIV Risk Score (DHRS) and the Behavioral Risk Screening Tool (BRST), as well as results of rapid HIV testing, if performed. Because HIV infection is a reportable disease, identifying information will be collected. While the final dataset will be stripped of identifiers prior to release for sharing, we believe that there remains a possibility of deductive disclosure of subjects with unusual characteristics. Thus, we will make data and associated documentation available to users only under a data-use agreement (DUA).
Supporting Information: Study Protocol
Time Frame: Data will become available after the main trial results have been reported/published. They will be available for a period of 10 years.
Access Criteria: Individuals who wish to access deidentified IPD must email the PI (Jason Haukoos) or Project Manager (Emily Caruso) with a description of the proposed analysis, outcomes of interest, and how results will be reported.

REFERENCES:
- [Derived] Haukoos JS, Lyons MS, Rothman RE, White DAE, Hopkins E, Bucossi M, Ruffner AH, Ancona RM, Hsieh YH, Peterson SC, Signer D, Toerper MF, Saheed M, Pfeil SK, Todorovic T, Al-Tayyib AA, Bradley-Springer L, Campbell JD, Gardner EM, Rowan SE, Sabel AL, Thrun MW; HIV TESTED Trial Investigators. Comparison of HIV Screening Strategies in the Emergency Department: A Randomized Clinical Trial. JAMA Netw Open. 2021 Jul 1;4(7):e2117763. doi: 10.1001/jamanetworkopen.2021.17763. PMID 34309668
- [Derived] Mohareb AM, Patel AV, Laeyendecker OB, Toerper MF, Signer D, Clarke WA, Kelen GD, Quinn TC, Haukoos JS, Rothman RE, Hsieh YH. The HIV Screening Cascade: Current Emergency Department-Based Screening Strategies Leave Many Patients With HIV Undiagnosed. J Acquir Immune Defic Syndr. 2021 May 1;87(1):e167-e169. doi: 10.1097/QAI.0000000000002609. No abstract available. PMID 33769768